CLINICAL TRIAL: NCT06792721
Title: EVALUATION OF CANCER RISK BY MEASUREMENT OF CIRCULATING MUTATIONAL BURDEN IN CARRIERS OF A GENETIC PREDISPOSITION
Brief Title: MEASUREMENT OF CIRCULATING MUTATION BURDEN
Acronym: cRISK
Status: Recruiting | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A02540-47
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Carcinoma; Genetic Predisposition to Cancer; BRCA Mutation; cfMB; Mutation Burden
Keywords: cfMB; predisposition to cancer; BRCA1; BRCA2; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for mutation Burden cfMB analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: participant with a hereditary predisposition linked to a BRCA1/2 mutation (case)
  Interventions: Genetic: Mutation Burden cfMB analysis
- Control group: participant not carrying a hereditary predisposition linked to a BRCA1/2 mutation (control) participant from the same sibling as the carrier participant (sister)
  Interventions: Genetic: Mutation Burden cfMB analysis

INTERVENTIONS:
Genetic: Mutation Burden cfMB analysis — Blood samples will be collected (one time only)

SUMMARY:
Cancer-free women with a hereditary predisposition to breast and/or ovarian cancer

DETAILED DESCRIPTION:
This proof-of-concept trial will be conducted with family members being monitored for a predisposition to breast and/or ovarian cancer linked to a BRCA1/2 gene mutation.

The study will be proposed to two sisters from the same sibling:

* one is a carrier of the genetic mutation
* and the other not,

Blood tests will evaluate the Mutation Burden cfMB

ELIGIBILITY:
Inclusion Criteria:

* Female participant
* Participant undergoing oncogenetic follow-up at the Centre François Baclesse
* Participant belonging to a pair of related biological siblings
* Within the sibling pair, one participant is a carrier of a hereditary predisposition linked to a BRCA1/2 mutation (case), and the other participant is not a carrier (control).
* Participant between 30 and 50 years of age
* Participant affiliated to a social security scheme
* Participant having given her consent to participate by signing an informed consent form prior to any specific study-related procedure.

Exclusion Criteria:

-

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participant is a carrier of a hereditary predisposition linked to a BRCA1/2 mutation (case), and the other participant (sister) is not a carrier (control).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the mutational burden in a person genetically predisposed to cancer with that of a non-predisposed relative | At the enrollment in the study (one point)
  Measurement and quantification of genomic signature on circulating DNA (mutational burden) derived from whole blood in a carrier of the genetic mutation and in her non-carrier first-degree relative.

SECONDARY OUTCOMES:
Mutation profiling, COSMIC-type signature generation | At the enrollment in the study (one point)
  Evaluate mutational signatures on circulating free DNA (cfDNA) in correlation with hereditary predisposition linked to the BRCA1 and BRCA2 genes
Identify and evaluate complementary or alternative molecular signatures | At the enrollment in the study (one point)
  Study of epigenetic biomarkers, such as circulating histone methylation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France, France

IPD SHARING:
Plan to Share IPD: No